CLINICAL TRIAL: NCT07108647
Title: In-Season Prevalence and Management of Hip and Groin Injuries in Competitive Athletes
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB25-0338
Record Dates: First submitted 2025-07-17; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Femoroacetabular Impingement Syndrome
Keywords: athletes; competitive; adolescent; young adult
MeSH Terms: conditions — Femoracetabular Impingement | interventions — Autogenic Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention (Experimental): Participants in the experimental arm will complete a 12-week, in-season progressive exercise program designed to improve hip strength, motor control, and function.
  Participants will complete a training session with a study trained clinician prior to beginning each respective phase of the program, either in person, or virtually per the participant preference.
  Participants will have the option to complete the intervention following a guided video for each phase, or on their own, at a location of their choosing, a minimum of three times per week.
  Interventions: Other: Progressive Hip Strengthening Program
- Time and Attention Control (Sham Comparator): Participants in the control arm will complete a 12-week, three-phase progressive muscle relaxation (PMR) program, adapted from the Jacobson method.
  Participants will complete a training session with a study trained clinician prior to beginning each respective phase of the program, either in person, or virtually per the participant preference.
  Participants will have the option to complete the intervention following a guided audio for each phase, at a location of their choosing, a minimum of three times per week.
  Interventions: Other: Progressive Muscle Relaxation

INTERVENTIONS:
Other: Progressive Hip Strengthening Program — This 12-week, in-season exercise intervention is designed for athletes with FAI syndrome and consists of three progressive phases.
  Phase 1 (Weeks 1-4): Focus on neuromuscular re-education and motor control using low-load exercises to improve hip and core activation, alignment, and stability.
  Phase 2 (Weeks 5-8): Targeted strengthening with increased load and movement complexity, emphasizing single-leg control, endurance, and pelvic stability.
  Phase 3 (Weeks 9-12): Integration of dynamic control, proprioception, and sport-specific movement patterns to support return to performance.
  Exercises target gluteus medius, gluteus maximus, core musculature, and functional movement systems. Participants complete the program >=3 times per week. Weekly questionnaires will monitor symptoms, adherence, and other management (e.g., physiotherapy).
  Arms: Exercise Intervention
Other: Progressive Muscle Relaxation — Participants in the time and attention control group will complete a 12-week, three-phase progressive muscle relaxation (PMR) program based on the Jacobson method. Phase 1 introduces isolated muscle tensing and relaxing to build awareness of muscle tension and promote body-mind connection. Phase 2 focuses on sequential relaxation of muscle groups, enhancing control and reducing stress. Phase 3 transitions to full-body relaxation through guided breathing and visualization techniques. Sessions are practiced 2-3 times per week using audio guides, with weekly check-ins from study staff. Symptom response, adherence, and participant experience are tracked throughout the season.
  Arms: Time and Attention Control

SUMMARY:
This study is focused on helping athletes with a common hip condition called femoroacetabular impingement (FAI) syndrome. FAI syndrome occurs when abnormal bone shapes around the hip joint cause friction during movement, leading to pain, reduced performance, and, over time, more serious injury. While this issue is well-studied in male professional athletes, little is known about how it affects female and collegiate athletes, or how to prevent it from worsening.

In this study, athletes diagnosed with FAI syndrome will participate in a 12-week in-season exercise program designed to reduce pain, improve hip strength and movement, and help prevent further injury-all while continuing their regular sports training.

Participants will be randomly assigned to either:

* An exercise group (receiving the intervention), or
* A time-and-attention control group (regular check-ins and education).

At the end of the study, the control group will have the option to access the exercise program.

The study will track changes in pain, physical performance, injury recurrence, and athlete satisfaction with the program. This research aims to improve how we manage hip injuries in athletes and help keep them active during the competitive season.

DETAILED DESCRIPTION:
Study Rationale Femoroacetabular impingement (FAI) syndrome is a common source of hip pain in athletes participating in cutting, pivoting, and high-impact sports such as soccer, basketball, ice hockey, and ringette. It is characterized by abnormal contact between the femoral head and acetabulum, which may lead to cartilage damage, labral tears, and early osteoarthritis. While research has primarily focused on male professional athletes, there is limited evidence regarding the early management of FAI in younger, female, and collegiate athletes.

Current management strategies often emphasize post-season rehabilitation or surgical interventions, limiting opportunities to explore conservative strategies that allow continued play during the competitive season. This randomized controlled trial (RCT) addresses that gap by evaluating a novel, in-season, 12-week exercise intervention designed to mitigate symptoms, maintain sport participation, and potentially delay or reduce long-term structural damage.

Study Objectives

1. Evaluate the feasibility of implementing an in-season, supervised exercise program in athletes with FAI syndrome.
2. Explore preliminary effectiveness signals on functional outcomes and symptom progression.

Study Design Participants diagnosed with FAI syndrome based on clinical evaluation and symptom history will be randomized to either the intervention or a time-and-attention control group. The intervention group will complete a structured neuromuscular and hip-specific rehabilitation program, while the control group receives educational support and a progressive mobility and recovery (PMR) option during the same 12-week period. Randomization ensures balanced comparison of feasibility and clinical endpoints.

Intervention Protocol

The 12-week intervention focuses on:

* hip and core strength (e.g., isometric and isotonic exercises targeting hip flexors, abductors, adductors, and gluteals)
* neuromuscular control (e.g., drills for dynamic stability, pelvic alignment, and functional control)
* functional progression (e.g., graded loading to meet game demands)

Participants complete the exercises a minimum of 3 times/week, and will be trained at the start of each phase in-person or remotely by a trained clinician. Exercise progression will occur after 4 weeks per phase. Compliance is monitored through weekly questionnaires.

Control Group Protocol: Time and Attention Control + PMR Option The control group will not participate in the structured exercise program but will receive supportive follow-up and access to a three-phase progressive muscle relaxation (PMR) program (audio guided). This design ensures time and engagement are balanced across groups.

The control group protocol includes:

* scheduled check-ins every 4 weeks with the research team for education and monitoring
* educational modules on injury prevention, load management, and hip health
* access to a guided three-phase PMR program

While participation in the PMR component is optional, it offers a low-intensity, restorative alternative without introducing strength training or neuromuscular drills that may overlap with the primary intervention. Control group participants are also offered the full exercise protocol following study completion.

Significance

This is one of the first studies to investigate an in-season, non-operative intervention for FAI syndrome in athletes during competitive play. It targets a high-risk group (female and collegiate athletes), with potential to:

* fill a critical gap in early-stage, conservative management of FAI syndrome
* inform future sport- and sex-specific injury prevention programs
* guide clinical decision-making regarding rehabilitation timing and delivery

Feasibility findings will guide future larger-scale studies, including refined criteria for participant selection, adherence support, and integration within team-based medical models.

ELIGIBILITY:
Inclusion Criteria:

* currently identifies as a "competitive athlete" based on the LTAD
* aged 14-40
* be free from any significant lower extremity injury (hip, groin, knee, ankle foot) in the past 6 months that resulted in >1 months of time loss or current inability to fully participate in sport at the time of baseline testing

If participants meet the above criteria, can be screened:

- completed bilateral hip screen, including imaging, and identified as having FAI syndrome with no degenerative joint changes (if meet the remaining criteria,

Exclusion Criteria:

* Are currently experiencing or recovering from a lower extremity injury that resulted in >1 month time lost within the past 6 months
* are pregnant or may become pregnant during the study (due to radiographic imaging exposure)
* * participants will be excluded from eligibility of RCT if they have evidence of moderate to severe osteoarthritis on imaging (Tönnis grade 2-3)

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of Agreement to Screening | up to 9 months - study time frame is 12 months, with the last participant able to enroll at month 9 to allow for 12 weeks of intervention
  the number of participants whom agree to be screened/the number of participants approached for recruitment
Eligibility Proportion | up to 9 months - study time frame is 12 months, with the last participant able to enroll at month 9 to allow for 12 weeks of intervention
  the number screened positive for inclusion (evidence of FAI syndrome)/number of participants who agreed to be screened (consented)
Consent Proportion | up to 9 months - study time frame is 12 months, with the last participant able to enroll at month 9 to allow for 12 weeks of intervention
  Number of participants screened positive and agreed to participate in intervention/number screened positive for inclusion
Randomization Proportion | up to 9 months - study time frame is 12 months, with the last participant able to enroll at month 9 to allow for 12 weeks of intervention
  The number of participants randomized/the number of participants screened positive and agreed to participate
Trial-Arm Selection Proportion | up to 9 months - study time frame is 12 months, with the last participant able to enroll at month 9 to allow for 12 weeks of intervention
  The number agreed to each trial arm after randomization/the number of participants randomized
Attrition Proportion | up to 9 months - study time frame is 12 months, with the last participant able to enroll at month 9 to allow for 12 weeks of intervention
  The number of participants who drop out of study/number of participants randomized in each arm

SECONDARY OUTCOMES:
International Hip Outcome Tool (iHOT-33) | 12 weeks
  The International Hip Outcome Tool (iHOT-33) is a 33-item patient-reported outcome measure designed to assess the health-related quality of life for young, active individuals with hip disorders. It focuses on how hip problems impact their daily activities, sports, work, and overall well-being. The iHOT-33 is a valuable tool for initial assessments, post-operative follow-ups, and clinical studies related to hip conditions.
Copenhagen Hip and Groin Outcome Tool (HAGOS) | 12 weeks
  Patient-reported questionnaire designed to assess the impact of hip and/or groin problems on physical function and quality of life in young to middle-aged, physically active individuals.
Make (Isometric) Strength Testing of the Hip | 12 weeks
  Strength measures in the hip (N/kg) performed in flexion, abduction, adduction. Measures will be performed pre and post intervention.
Passive Range of Motion | 12 weeks
  Range of motion in degrees at the hip joint in flexion, internal rotation, abduction. Performed pre and post intervention.
Special Test Findings | 12 weeks
  Positive or negative findings on special tests in the hip which reproduce the pain of an injury (out of a maximum of 3). Performed pre and post intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Emery, PT, PhD, Principal Investigator — Sport Injury Prevention Research Centre, Chair

IPD SHARING:
Plan to Share IPD: No